CLINICAL TRIAL: NCT05013580
Title: The "Open Wound Bone Augmentation Concept" with Amnion-Chorion Membrane: a Randomized Controlled Trial
Brief Title: The "Open Wound Bone Augmentation Concept" with Amnion-Chorion Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Muhammad Saleh, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00161016
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-09

CONDITIONS: Horizontal Ridge Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open Wound (Experimental): After horizontal bone grafting, the wound where the graft was attached to the bone will be filled with a type of tissue (the amnion-chorion membrane) taken from a placenta and will be left partially open to heal.
  Interventions: Procedure: Guided bone regeneration (GBR)
- Closed Wound (Active Comparator): After horizontal bone grafting, the wound where the graft was attached to the bone will be filled with collagen tissue and stitched closed while it heals.
  Interventions: Procedure: Guided bone regeneration (GBR)

INTERVENTIONS:
Procedure: Guided bone regeneration (GBR) — Bone grafts will be placed in the patient's jawbone, along with a membrane to cover the bone grafts. A horizontal incision over the edentulous ridge crest will be made along with vertical incisions if indicated. Buccal and lingual full thickness mucoperiosteal flaps will be reflected to expose the alveolar bone. Intra-marrow penetration (decortication of the alveolar bone to increase vascular supply to the bone grafts) at the surgical site alveolar bone will be made with a high-speed hand piece and diamond bur. Bone allograft material will be placed to fill the alveolar bone defect. The bone graft will then be covered with a membrane and secured with sutures.
  Other Names: Horizontal bone augmentation (HBA)

SUMMARY:
The purpose of this study is to compare two bone graft wound healing techniques; an open wound healing approach versus the standard closed wound healing approach.

DETAILED DESCRIPTION:
Open wound healing approach (experimental technique): the wound where the graft was attached to the bone will be filled with a type of tissue (the amnion-chorion membrane) taken from a placenta (the tissue sac that surrounds an embryo) and will be left partially open to heal.

Closed wound healing approach (standard technique): the wound where the graft was attached to the bone will be filled with collagen tissue (processed bone grafts from donors) and stitched closed while it heals.

20 patients needing more bone before placing a dental implant will be recruited for this trial. Patients will be randomized to either the test (open wound healing approach) or control (closed wound healing approach) group.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age
* Be missing 1 to 2 back teeth in the lower jaw for at least three months
* Need horizontal bone ridge augmentation (gain width of the bone) prior to implant placement, determined clinically and radiographically
* Have enough bone height at the site

Exclusion Criteria:

* Currently smoke more than 10 cigarettes a day (self-reported)
* Have any medical conditions or jaw pathology that we decide might influence the outcome of the study
* Are pregnant or are lactating (self-reported)
* Have unstable periodontal disease or other dental infection
* Have poor oral hygiene
* Have any clinical conditions that make the subject unsuitable for bone graft surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Ridge width changes | 6 months
  Radiographic changes of the ridge width based on cone-beam computed tomography (CBCT) scan measurements

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Saleh, BDS, MSD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No